CLINICAL TRIAL: NCT00474864
Title: A Double-Blind, Placebo-Controlled, Parallel Study To Evaluate The Effects Of GW856553 On Endothelial Function/Vascular Compliance In Subjects With Dyslipidaemia.
Brief Title: Study To Evaluate The Effects Of GW856553 On Endothelial Function/Vascular Compliance In Subjects With Dyslipidaemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PM1108357
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Subjects; Dyslipidaemias; Dyslipidaemia
Keywords: Endothelial Function,; vascular compliance,; atherosclerosis
MeSH Terms: conditions — Dyslipidemias; Atherosclerosis | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW856553

SUMMARY:
The rationale for this study is to determine whether GW856553 (7.5mg BD for 28 days) has an effect on endothelial function in dyslipidaemic subjects as assessed by venous occlusion plethysmography using brachial artery acetylcholine infusion. This will establish consistency with preclinical findings, as well as confirm a physiologic human response at the current safe maximal dose. Safety (specifically serum liver function testing) and tolerability will also be evaluated in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and females between 18 and 75 years of age, inclusive.
* To be eligible, female subjects must have a negative pregnancy test (i.e. Urine or serum β-hCG (for females) and be of:

  * non-childbearing potential (i.e. physiologically incapable of becoming pregnant). This includes any female who is post-menopausal.

OR

* childbearing potential and agree to commit to one of the protocol-approved methods of contraception.

  * Body weight > 50 kg and body mass index (BMI) between 19 and 32kg/m2
  * Subjects with high LDLc levels, as per NCEP ATPIII criteria:fasting LDLc level > 4.1 mmol/L (160 mg/dL), inclusive. Fasting TG level should be < 4.5mmol/L (400 mg/dL)
  * A signed and dated written informed consent prior to admission to the study
  * The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

The following criteria must apply only for subjects undergoing FDG-PET/CT and MRI

* All diabetics will be excluded from the scanning sub-study involving MRI and FDGPET/CT.
* Subjects will be excluded who have previously participated in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden (a significant radiation burden being defined as ICRP category IIb or above: No more than 10 mSv effective radiation dose in addition to natural background radiation, in the previous 3 years including the dose from this study). Given the planned administration of 10 mSv in this study, any subjects who have been exposed to ionizing radiation above background levels, for example as a result of their work with radiation as category A (classified) workers, will be excluded
* Adult males and females between 50 and 75 years of age, inclusive.
* Women must be of non-childbearing potential [i.e. either postmenopausal or documented hysterectomy - tubal ligation is not sufficient]. To be eligible, female subjects must have a negative pregnancy test (i.e. serum beta hCG test) and be of non-childbearing potential (i.e. physiologically incapable of becoming pregnant). This includes any female who is post-menopausal. All diabetics will be excluded from the scanning sub-study involving MRI and FDG-PET/CT.
* Contraindication to MRI scanning (as assessed by local MRI safety questionnaire) which includes but not limited to:
* Intracranial aneurysm clips (except Sugita) with an appropriate operative conformation,
* History of intra- orbital metal fragments that have not been removed by an MD,
* Pacemakers and non-MR compatible heart valves,
* Inner ear implants,
* History of claustrophobia in MR.
* Is unable to lie comfortably on a bed inside a PET camera with their head in the field of view for at least 60 minutes as assessed by physical examination and medical history (e.g. back pain, arthritis).

The following criteria apply only for healthy control subjects

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Healthy adult male between 18 and 75 years of age, inclusive.
* Body weight > 50 kg and body mass index (BMI) between 19 and 32kg/m2
* A signed and dated written informed consent prior to admission to the study
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Blood pressure should be <=140 mmHg systolic and/or <=90mmHg diastolic)
* Subjects with LDLc, < 2.6 mmol/L (100 mg/dL). Fasting TG level should be <1.7mmol/L (150 mg/dL); HDLc > 1.0 mmol/L (40mg/dL)
* Non-smokers

Exclusion Criteria:

* History of symptomatic coronary artery disease, stroke, or other known atherosclerotic disease.
* Subjects who are current smokers and require a cigarette within 30 minutes after they wake in the morning, or cannot abstain from smoking for approximately 5 hours.
* History of chronic viral hepatitis (including presence of hepatitis B surface antigen or hepatitis C antibody), or other chronic hepatic disorders.
* History of increased liver function tests (ALT, AST) due to acute or chronic liver conditions, above the upper limit of normal in the past 6 months and/or liver function tests (bilirubin, ALT, AST) above the upper limit of normal at Screening.
* Renal impairment with creatinine clearance of <50 ml/min at screening, or history of kidney transplant or history of contrast nephropathy.
* Current inadequately controlled hypertension (blood pressure >180 mmHg systolic and/or >100mmHg diastolic) or any subject who has experienced a modified regimen of antihypertensive medication within 6 weeks prior to first dose of study medication, or any subject who is likely to commence treatment of a hypertensive medication
* Current poorly controlled diabetes mellitus, defined as HbA1c >10% at Screen.
* History of heart failure defined as NYHA class II - IV or those with known severe LV dysfunction (EF<30%) regardless of symptomatic status
* History of malignancy within the past 5 years, other than non-melanoma skin cancer.
* Current life-threatening condition other than vascular disease (e.g., very severe chronic airways disease, HIV positive, life-threatening arrhythmias) that may prevent a subject from completing the study.
* Alcohol or drug abuse within the past 6 months.
* Previous exposure to GW856553.
* Use of an investigational device or investigational drug within 30 days or 5 half-lives (whichever is the longer) preceding the first dose of study medication.
* Subjects who will commence or who are likely to commence treatment with oral intranasal or topical corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs) (other than aspirin), PPARγ agonists (e.g. rosiglitazone), sulfonylureas, insulin, fibrates, niacin, ACEI, ARBs, nitrates, HRT, etc from screening until study completion.
* Any non-stable dosing of ongoing medication regimens (as noted above (#14)) throughout the study trial.
* Any subject that is likely to commence statin treatment from screening until the final follow up visit. Any subjects currently receiving treatment with statins must be able to washout from the statin for 28 days prior to first dose of study medication.
* The subject has a three month prior history of regular alcohol consumption exceeding an average weekly intake of > 28 units (or an average daily intake of greater than 3 units) for males, or an average weekly intake of > 21 units (or an average daily intake of greater than 2 units) for females or a positive alcohol breath test at the screening visit
* A positive urine test for drugs of abuse (not related to known medications the subject is taking, ie, codeine for pain management) or alcohol at screening or prior to study medication administration.
* Any other subject whom the Investigator deems unsuitable for the study (e.g., due to either medical reasons, laboratory abnormalities, expected study medication non-compliance, or subject's unwillingness to comply with all study-related study procedures).
* Subjects with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with chronic inflammation (e.g. Inflammatory Bowel Disease).
* Subjects with chronic infections such as gingivitis, periodontitis, prostatitis, gastritis, and urinary tract infections, or any active diseases, including active tuberculosis or a history of active tuberculosis.
* Subjects with any acute infection, symptoms suggestive of sinusitis, or significant trauma (burns, fractures).
* Subjects who have donated more than 500 mL of blood within 56 days prior to the study medication administration.
* History of myopathy or rhabdomyolysis.
* QTc interval >450 msec
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women; or an unwillingness of the subject to use contraceptive methods defined in the protocol from the time of the first dose of the study medication until 3 months after administration of last dose of study medication.
* Pregnant or nursing women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow ratio measured at baseline and day 28. | at baseline and day 28.

SECONDARY OUTCOMES:
Forearm blood flow ratio at (baseline and day28). Augmentation Index(baseline and day28). Pulse wave velocity (baseline and day28). pHSP-27 levels (baseline and day28). | baseline and day28
Safety and tolerability parameters (weekly) | weekly
Measurement of total and phosphorylated heat shock protein-27 (pHSP-27) levels in sorbitol induced whole blood cells of patients with dyslipidaemia
Safety and tolerability parameters, including physical examination, blood pressure, heart rate, 12-lead electrocardiograms (ECGs), clinical laboratory tests, and adverse events reporting

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - GSK Investigational Site, London, London
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Cardiff

REFERENCES:
- [Derived] Cheriyan J, Webb AJ, Sarov-Blat L, Elkhawad M, Wallace SM, Maki-Petaja KM, Collier DJ, Morgan J, Fang Z, Willette RN, Lepore JJ, Cockcroft JR, Sprecher DL, Wilkinson IB. Inhibition of p38 mitogen-activated protein kinase improves nitric oxide-mediated vasodilatation and reduces inflammation in hypercholesterolemia. Circulation. 2011 Feb 8;123(5):515-23. doi: 10.1161/CIRCULATIONAHA.110.971986. Epub 2011 Jan 24. PMID 21262998